CLINICAL TRIAL: NCT05580627
Title: Relationships Education, Financial Resources, & Anger Management Essentials (REFRAME)
Brief Title: Evaluation Exploring How Course Modality Influences the Effectiveness of the R3 Academy for Couples
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healthy Relationships California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 90ZB0026
Record Dates: First submitted 2022-09-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Program Modality
Keywords: couple relationship education; modality; evaluation; couple; comparison; propensity score matching; live; in-person; livestream; online
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: In our quasi-experimental design, we allow participants to select whether they want to participate in a live or livestream program modality. The couples curriculum is the same for both, only the mode of delivery is different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Livestream Modality (Experimental): The livestream modality is considered the treatment group for the purpose of this quasi-experimental study.
  Interventions: Other: Livestream Modality (treatment)
- Live Modality (Experimental): The live modality is considered the control group for the purpose of this quasi-experimental study.
  Interventions: Other: Live Modality (control)

INTERVENTIONS:
Other: Livestream Modality (treatment) — For this evaluation, the livestream modality is considered the treatment group.
  Arms: Livestream Modality
Other: Live Modality (control) — For this evaluation, the live modality is considered the control group.
  Arms: Live Modality

SUMMARY:
The REFRAME project is designed to offer the R3 Academy for Couples, a robust 24-hour program, to married adults ages 18 and over in the state of California. The R3 Academy is an evidence-based couple relationship education curriculum that helps couples strengthen their relationships with their child, with their spouse, and at work. The program also includes two evidence-based components that address economic stability and an innovative approach to Case Management that fosters client self-direction. The R3 Academy curricula will be delivered in both English and Spanish through two modalities: 1) live classes and 2) livestream classes via a video conferencing platform. The Local Evaluation will examine how modality, or in other words attending a live class versus a livestream class, influences the effectiveness of R3 Academy for Couples program when it comes to changes in couples' marital/relationship satisfaction, conflict management, support and affection, and commitment. The question of modality is a timely one. In the COVID-19 era, many programs have become exclusively online-but the potential impact on effectiveness is not well known. We address this issue by considering the impact on four relationship outcomes: marital/relationship satisfaction, conflict management, support and affection, and commitment. Moreover, one issue that many programs report is that couples have great difficulty finding time to be engaged in regularly scheduled, live, in-person classes. Our study will provide evidence about how the availability of materials in alternative formats, that may allow more couples to be involved and reduce issues around the ability to participate, may influence the efficacy of those programs.

RQ1: How do live in-person (control) and online livestream (treatment) Marriage and Relationship Education (MRE) workshops compare on marital/relationship satisfaction outcomes immediately after program completion? RQ2: How do live in-person and online livestream MRE workshops compare on conflict management outcomes immediately after program completion? RQ3: How do live in-person and online livestream MRE workshops compare on support and affection outcomes immediately after program completion? RQ4: How do live in-person and online livestream MRE workshops compare on commitment outcomes immediately after program completion? RQ5: Do program effects last beyond program completion?

DETAILED DESCRIPTION:
Couples in this study are required to take an Eligibility survey. If they meet the required eligibility criteria, the survey will gather further information including screening factors associated with domestic violence and child maltreatment that, if checked, will be flagged for further assessment by personal contact with our Case Management Supervisor. This form will also enable the registrant to identify which class format he or she wishes to attend-a live R3 Academy or a livestream workshop via a video conferencing platform. For the purpose of this study, the live or in-person modality is considered the control group and the livestream workshop is considered the treatment group. The R3 Academy curriculum is the same for each group, only the modality of curriculum delivery is different. Courses are a total of 24 hours that stretch across 12 sessions. Incentives for program completion include a $50 gift card that is offered to those who complete at least 90% of the program. In addition to the Eligibility survey, participants are asked to take a pre-survey before starting the class, a post-survey immediately following class completion, and a 4-month follow-up survey. If participants complete all three surveys they are eligible for an additional $25 gift card which they can receive even if they did not reach 90% completion.

As stated previously, entry into treatment or control groups is determined at enrollment. At the time of the impact analysis, propensity score matching (PSM) comparison groups will be formed-this statistical analysis will match up similar participants from each group to allow for comparison across conditions. PSM allows researchers to estimate differences between treatment and control groups in non-randomized samples. PSM will allow us to directly compare matched cases-meaning that the treatment and control groups will have a similar distribution of sociodemographic and sociocultural characteristics. This allows us to consider how outcomes vary between treatment and control groups, while accounting for the potential self-selection into different program groups. Participants will be matched across multiple metrics, including: racial/ethnic identity, sex/gender, income, education level, language of instruction, number of children, employment status, age, marital status, residential status, child sex, and child age. As clients may choose one program delivery modality over another due to work, childcare availability, or time, measures will be included for work schedule, availability of social support, work flexibility, and work-family stress.

ELIGIBILITY:
Inclusion Criteria:

* Adult over the age of 18 living in California and applying with their romantic partner

Exclusion Criteria:

* Domestic violence or child maltreatment is detected
* Active drug use
* Undiagnosed or untreated mental illness
* Anger management issues
* Pending legal action

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Marital/Relationships Satisfaction after program completion and 4 months following program completion | Data is collected at three time points: (1) before attending the class, (2) immediately after class completion, and (3) 4 months after course completion.
  Single item inquiring how satisfied the individual is with their relationships. Responses are given on a Likert scale from 1=very satisfied and 3=not satisfied.
Change in Conflict Management after program completion and 4 months following program completion | Data is collected at three time points: (1) before attending the class, (2) immediately after class completion, and (3) 4 months after course completion.
  2 subscales and one single question exploring difficulty with working out differences, respect during disagreements, and satisfaction with conflict resolution. The first 2 are multiple item scales presented on a scales inquiring how frequently example interaction occur with responses given on a Likert scale ranging from 1=Never to 4=Often. Satisfaction with conflict resolution is based on a single question asking how satisfied the individual is with their conflict management. Responses are given on a Likert scale ranging from 1=Very satisfied to 3=Not at all satisfied.
Change in Partner Support after program completion and 4 months following program completion | Data is collected at three time points: (1) before attending the class, (2) immediately after class completion, and (3) 4 months after course completion.
  This is based on a 5-item measure inquiring how much participants agree or disagree with a list of statements related to their partner's supportiveness. Responses are given on a Likert scale ranging from 1=Strongly agree to 4=Strongly disagree.
Change in Relationship Commitment after program completion and 4 months following program completion | Data is collected at three time points: (1) before attending the class, (2) immediately after class completion, and (3) 4 months after course completion.
  This outcome is measured with a single item inquiring how much participants agree or disagree with the statement: I view our relationships as being life-long. Responses are given on a Likert scale ranging from 1=Strongly agree to 4=Strongly disagree.
Change in Partner Affection after program completion and 4 months following program completion | Data is collected at three time points: (1) before attending the class, (2) immediately after class completion, and (3) 4 months after course completion.
  This scale explored how frequently participants experience a list of 3 interactions with their partners. Responses are given on a Likert scale ranging from 1=Almost every day to 4=Less often.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Shafer, PhD, Principal Investigator — Brigham Young University; Jason Krafsky, Study Director — Healthy Relationships California; Patty Howell, Study Chair — Healthy Relationships California; Dyann Collins, Study Chair — Healthy Relationships California
Locations (1):
- Healthy Relationships California, Leucadia, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be archived with the Inter-university Consortium for Political and Social Research (ICPSR) after we complete our research. The data will not include the participant's name, address, date of birth, phone number, or any other personal information or ID numbers that could identify the participant. Archiving this data provides other researchers with the opportunity to learn about how relationship education benefits people. Information about data archival will be provided on the consent form.